CLINICAL TRIAL: NCT02013804
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI0680 (AMP-514) in Subjects With Advanced Malignancies
Brief Title: A Phase 1 Multicenter Open-label Study to Evaluate the Safety Tolerability and PK of MEDI0680 (AMP-514) in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP-514-01; D6020C00002 (AMP-514-01) (Other: MedImmune)
Record Dates: First submitted 2013-12-12; First posted 2013-12-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose arms (Experimental): Dose Escalation
  Interventions: Drug: MEDI0680 (AMP-514)

INTERVENTIONS:
Drug: MEDI0680 (AMP-514) — Study has planned dose escalation cohorts

SUMMARY:
This is a multicenter, open label, first-in-human dose-escalation study of MEDI0680 (AMP-514) to evaluate the safety, tolerability, PK, immunogenicity (IM), and antitumor activity in adult subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at time of study entry
2. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act [HIPAA] in the USA) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
3. Histologically- or cytologically-confirmed melanoma or clear-cell RCC that are refractory to standard therapy or for which no standard therapy exists

   1. Subjects must have failed, be intolerant to, or be ineligible for any potentially curative approved treatment, irrespective of line of therapy
   2. No more than 3 prior lines of therapy
4. At least 1 measurable lesion per RECIST v1.1; subjects whose only measurable lesion is a lymph node will be excluded
5. Eastern Cooperative Oncology Group performance score of 0 or 1
6. For all tumor types, adequate organ and marrow function, as defined below:

   1. Hemoglobin ³ 9.0 g/dL within first 2 weeks prior to first dose of MEDI0680 (AMP-514)
   2. Absolute neutrophil count (ANC) ³ 1.5 × 109/L (1,500/mm3)
   3. Platelet count ³ 100 × 109/L (100,000/mm3)
   4. Total bilirubin ≤ 1.5 × ULN except subjects with documented Gilbert's syndrome (> 3 × ULN) or liver metastasis, who must have a baseline total bilirubin ≤ 3.0 mg/
   5. Alanine aminotransferase and AST ≤ 2.5 × ULN; for subjects with hepatic metastases, ALT and AST ≤ 5 × ULN
   6. Serum creatinine ≤ 1.5 × ULN OR calculated creatinine clearance (CrCl) or 24-hour urine CrCl ≥ 50 mL/minute ▪ Cockcroft-Gault formula will be used to calculate CrCl; 24-hour urine CrCl will be derived using the measured creatinine clearance formula
7. Prior treatment toxicities must be ≤ Grade 1

Exclusion Criteria:

1. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
2. Receipt of any BRAF inhibitor (in metastatic melanoma), or investigational anticancer therapy within 4 weeks prior to the first dose of MEDI0680 (AMP-514)
3. Prior exposure to immunotherapy, such as, but not limited to, other anti-CTLA-4, anti-PD-1, or anti-PD-L1 antibodies, excluding therapeutic cancer vaccines
4. Major surgery (as defined by the investigator) within 4 weeks prior to first dose of MEDI0680 (AMP-514) or still recovering from prior surgery
5. Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured
6. Prior allogeneic or autologous bone marrow or organ transplantation that requires use of immunosuppressives
7. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v4.03 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by MEDI0680 (AMP-514) may be included (eg, hearing loss) after consultation with the MedImmune medical monitor
8. Active or prior documented autoimmune disease within the past 2 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability; define Maximum Tolerated dose | 1 year
  The primary objectives are to assess the safety and tolerability of multiple doses of MEDI0680 (AMP-514) and define the maximum tolerated dose (MTD) or highest protocol-defined dose of MEDI0680 (AMP-514) in the absence of exceeding the MTD.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, New Haven, Connecticut
  - Research Site, Detroit, Michigan
  - Research Site, The Bronx, New York
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

REFERENCES:
- [Derived] Naing A, Infante J, Goel S, Burris H, Black C, Marshall S, Achour I, Barbee S, May R, Morehouse C, Pollizzi K, Song X, Steele K, Elgeioushi N, Walcott F, Karakunnel J, LoRusso P, Weise A, Eder J, Curti B, Oberst M. Anti-PD-1 monoclonal antibody MEDI0680 in a phase I study of patients with advanced solid malignancies. J Immunother Cancer. 2019 Aug 22;7(1):225. doi: 10.1186/s40425-019-0665-2. PMID 31439037
- [Derived] Borch TH, Donia M, Andersen MH, Svane IM. Reorienting the immune system in the treatment of cancer by using anti-PD-1 and anti-PD-L1 antibodies. Drug Discov Today. 2015 Sep;20(9):1127-34. doi: 10.1016/j.drudis.2015.07.003. Epub 2015 Jul 17. PMID 26189934